CLINICAL TRIAL: NCT02688049
Title: The Efficacy and Safety of NeuroRegen Scaffold™ Combined With Mesenchymal Stem Cells or Neural Stem Cells for Chronic Spinal Cord Injury Repair
Brief Title: NeuroRegen Scaffold™ Combined With Stem Cells for Chronic Spinal Cord Injury Repair
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chinese Academy of Sciences (Other Government)
Collaborators: Affiliated Hospital of Logistics University of CAPF (Other)
Responsible Party: Principal Investigator, Jianwu Dai, Principal Investigator of Regenerative Medicine Laboratory, Institute of Genetics and Developmental Biology, CAS, Chinese Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAS-XDA-MNSCI/IGDB
Record Dates: First submitted 2016-02-06; First posted 2016-02-23 (Estimated); Last update posted 2020-12-23 (Actual); Status verified 2016-02

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NeuroRegen scaffold/mesenchymal stem cells transplantation (Experimental): Patients receive NeuroRegen scaffold with mesenchymal stem cells transplantation after spinal cord injury.
  Interventions: Biological: NeuroRegen scaffold/mesenchymal stem cells transplantation
- NeuroRegen scaffold/neural stem cells transplantation (Experimental): Patients receive NeuroRegen scaffold with neural stem cells transplantation after spinal cord injury.
  Interventions: Biological: NeuroRegen scaffold/neural stem cells transplantation

INTERVENTIONS:
Biological: NeuroRegen scaffold/mesenchymal stem cells transplantation — Patients with chronic SCI (ASIA grade A) will receive NeuroRegen Scaffold with 10 million mesenchymal stem cells transplantation after localized scars cleared and after surgery patients will undergo a comprehensive rehabilitation, psychological and nutritional measures.
  Arms: NeuroRegen scaffold/mesenchymal stem cells transplantation
Biological: NeuroRegen scaffold/neural stem cells transplantation — Patients with chronic SCI (ASIA grade A) will receive NeuroRegen Scaffold with 10 million neural stem cells transplantation after localized scars cleared and after surgery patients will undergo a comprehensive rehabilitation, psychological and nutritional measures.
  Arms: NeuroRegen scaffold/neural stem cells transplantation

SUMMARY:
The purpose of this study is to assess the efficacy and safety of mesenchymal stem cells or neural stem cells combined with NeuroRegen scaffold transplantation in patients with spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18-65 years old.
2. Completely spinal cord injury at the cervical and thoracic level (C5-T12).
3. Classification ASIA A with no significant further improvement.
4. Patients signed informed consent.
5. Ability and willingness to regular visit to hospital and follow up during the protocol Procedures.

Exclusion Criteria:

1. A current diagnosis of any primary diseases affecting limb functions (e.g., trauma, infection, tumors, congenital malformations, peripheral muscular dystrophy, Huntington's disease, Parkinson's disease).
2. Serious complications (e.g., hydronephrosis due to renal insufficiency, severe bedsores (Ⅲ° above), lower extremity venous thrombosis, severe myositis ossificans).
3. History of life threatening allergic or immune-mediated reaction.
4. Clinically significant abnormalities in routine laboratory examinations (hematology, electrolytes, biochemistry, liver and kidney function tests, urinanalysis).
5. History of mental illness or suicide risk, with a history of epilepsy or other central nervous system disorders.
6. Severe arrhythmias (e.g., ventricular tachycardia, frequent superventricular tachycardia, atrial fibrillation, and atrial flutter) or cardiac degree II or above conduction abnormalities displayed via 12-lead ECG.
7. Lactating and pregnant woman.
8. Alcohol drug abuse /dependence.
9. Participated in any other clinical trials within 3 months before the enrollment.
10. A drug or treatment known to cause effect on the central nervous system during the past four weeks.
11. A drug or treatment known to cause major organ system toxicity during the past four weeks.
12. Poor compliance, difficult to complete the study.
13. Any other conditions that might increase the risk of subjects or interfere with the clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-01; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Improvements in ASIA (American Spinal Injury Association) Impairment Scale | 24 months
Improvements in Somatosensory Evoked Potentials (SSEP) | 24 months
Improvements in Motor Evoked Potentials (MEP) | 24 months

SECONDARY OUTCOMES:
Improvements in Independence Measures | 1, 3, 6, 12, 18 and 24 months
  Functional Independence Measure (FIM) will be assessed before and after surgery.
Changes at the transplantation site in spinal cord by Magnetic Resonance Imaging (MRI) | 1, 3, 6, 12, 18 and 24 months
  The MRI at the transplantation site will be assessed before and after transplantation.
Improvements in Urinary and Bowel Function | 1, 3, 6, 12, 18 and 24 months
  The ability to feel and control urination and bowel will be assessed based on bladder pressure monitory before and after surgery.
Safety and Tolerability assessed by Adverse Events | Up to 6 months
  Proportion of patients with postoperative infections and serious adverse events (SAEs) will be assessed by long term follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Jianwu Dai, Ph.D, Principal Investigator — Chinese Academy of Sciences
Locations (1):
- Affiliated Hospital of Logistics Universtiy of CAPF, Tianjin, China